CLINICAL TRIAL: NCT02513251
Title: Validation of the Traditional Chinese-Cantonese Version of Short Form McGill Pain Questionnaire (C-SF-MPQ-2)
Brief Title: Chinese-Cantonese Version of Short Form McGill Pain Questionnaire Validation
Status: Completed | Type: Observational
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. Chi-Wai Cheung, Clinical Associate Professor, The University of Hong Kong
Other Study IDs: UW15-013
Record Dates: First submitted 2015-07-29; First posted 2015-07-31 (Estimated); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Chronic Pain
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Case group: Chronic pain patient
  Interventions: Other: Chronic pain

INTERVENTIONS:
Other: Chronic pain — Chronic pain patients would complete the Traditional Chinese-Cantonese version of Short Form McGill Pain Questionnaire

SUMMARY:
Pain is defined as "An unpleasant sensory and emotional experience associated with actual or potential tissue damage, or described in terms of such damage." In particular, chronic pain has significant impact on health care cost and socio-economic aspects of the society. It is clear that the development of effective chronic pain management is paramount in reducing the significant socio-economic burden of this common healthcare problem.

One of the difficulties in measuring outcomes in chronic pain patients is the subjective nature of pain. The McGill Pain Questionnaire (MPQ) was developed in 1975 with the aim of quantifying the subjective pain experiences of patients. Since then it has become one of the major assessment tools in evaluation of chronic pain patients during the course of treatments. The Short Form McGill Pain Questionnaire (SF-MPQ) developed in 1987 has further refined pain descriptors into "sensory" and "affective" domains, and incorporating the Visual Analog Scale (VAS) for easier administration in hospitals and clinics. The validity and reliability of both the original English and translated versions of MPQ and SF-MPQ have been well demonstrated. The latest version of Short Form McGill Pain Questionnaire (SF-MPQ-2) included descriptive terms for neuropathic pain which expanded the scope of coverage on chronic neuropathic pain patients. It has also been evaluated in cancer pain patients. Translated versions of SF-MPQ-2 showed good reliability and validity. Therefore the investigators devised this study to (1) translate SF-MPQ-2 into Traditional Chinese-Cantonese (C-SF-MPQ-2) suitable for use in Hong Kong patients, (2) examine the validity, reliability and psychometric properties of this translated version in Hong Kong patients.

DETAILED DESCRIPTION:
Objectives of this trial

1. To validate the C-SF-MPQ-2 among chronic pain patients in Hong Kong.
2. To evaluate the validity, reliability and psychometric properties of the C-SF-MPQ-2 as an assessment tool for measuring pain.

Trial design Prospective non-randomized trial with self-administered questionnaire in chronic pain patients.

Methods The study will be carried out in 2 phases (I and II). Phase I refers to the translation process and phase II refers to the validation process.

Since this study will be carried out at 2 pain centres (Hong Kong West Cluster Pain Management Centre and Kowloon East Cluster Pain Management Centre), approvals from Ethics Committee of Hong Kong West Cluster and Kowloon East Cluster will be obtained.

(I) Translation of the original English version of SF-MPQ-2 into Traditional Chinese-Cantonese version (C-SF-MPQ-2) Forward translation shall be done by one pain specialist and one lay person with linguistic background. Both shall be native Chinese-Cantonese speaker with proficiency in English. Each translator shall produce a translated version independently. Afterwards the principle investigator will co-ordinate with both translators to come up with one commonly agreed translated version (version 1).

Backward translation shall be done by one pain specialist who is a native English speaker with proficiency in Chinese-Cantonese (version 2). This will be compared to the original questionnaire. The principle investigator will discuss with all the translators on any discrepancy between version 2 and the original version and make necessary adjustments to version 1 to produce a revised version (version 3).

The translated version 3 will then be tested on 5 randomly selected chronic pain patients from both pain management centres. They shall be native Chinese-Cantonese speakers. Consent will be obtained beforehand. An interviewer will inquire whether patients have any difficulty on completing the questionnaire or have any suggestions with regard to the translated terms. Any adjustments shall be made after receiving feedback from the interviewer to produce the finalized version (C-SF-MPQ-2).

(II) Validation of C-SF-MPQ-2 A total of 220 chronic pain patients will be recruited for the process of validation. After obtaining consent, basic demographic information including age, sex, pain diagnosis and duration, education level, co-existing medical problems and employment status will be recorded. The C-SF-MPQ-2 will then be administered to patients. For the construct validity, the Chinese versions of Medical Outcome Study Short Form 36 (SF-36), ID-Pain and Pain Catastrophizing Scale (PCS) will be administered at the same time. For the test-retest reliability, the C-SF-MPQ-2 will be administered again after 2 weeks at the pain management centres during which patients should not receive any alternation in their pain management or intervention. Patients' data privacy and confidentiality will be ensured during the entire process of study.

ELIGIBILITY:
Inclusion Criteria:

* Native Chinese-Cantonese speaker
* Aged 18 or above
* Presence of chronic pain for more than 3 months
* Able to understand, read and write Traditional Chinese
* Mentally capable to give informed written consent
* Ability to complete the questionnaires

Exclusion Criteria:

* Non-native Chinese-Cantonese speaker
* Aged below 18
* Unable to read or write Traditional Chinese
* Presence of chronic pain for less than 3 months
* Mentally incapable to give informed written consent
* Unable to complete the questionnaires
* Patients who require active pain treatment and / or intervention within 2 weeks after the initial consultation
* Voluntary withdrawal from study at any stage

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Chronic pain patients from the Pain Clinic in Queen Mary Hospital
Sampling Method: Non-Probability Sample
Enrollment: 241 (Actual)
Dates: Start 2015-07-31 (Actual); Primary Completion 2021-05-31 (Actual); Study Completion 2023-07-31 (Actual)

PRIMARY OUTCOMES:
C-SF-MPQ-2 score | 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Chi Wai Cheung, MBBS, MD, Principal Investigator — The University of Hong Kong
Locations (1):
- Deaprtment of Anaesthesiology, The University of Hong Kong, Hong Kong, China